CLINICAL TRIAL: NCT05341050
Title: This Study is a Multicenter, Single-arm, Prospective Study to Evaluate the Efficacy and Safety of Drug Discontinuation After Dose Reduction in Ph+CML-CP Patients Threated With 2G-TKI.
Brief Title: A Study on the Withdrawal of Second-generation Tyrosine Kinase Inhibitors After Dose Reduction in Patients With CML
Status: Recruiting | Type: Observational
Sponsor: xuna (Other)
Responsible Party: Sponsor-Investigator, xuna, Associate chief physician, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Other Study IDs: TKIs-cml
Record Dates: First submitted 2022-04-09; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: MMR on 12 Month

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with Ph+ CML-CP
  Interventions: Drug: TKI

INTERVENTIONS:
Drug: TKI — halve dose of 2G-TKI for 12 months and then withdrawal for 12 months

SUMMARY:
patients with Ph+ CML-CP who have been treated with second-generation TKIs (nilotinib, dasatinib) for at least 3 years and maintains MMR for at least 2 years, continue to be treated with halved dose for 12 months, and then stop for 12 months.

DETAILED DESCRIPTION:
1.Patients with Ph+ CML-CP who have been treated with second-generation TKIs (nilotinib, dasatinib) for at least 3 years and maintains MMR for at least 2 years.

2。During the TKI reduction phase, the peripheral blood BCR/ABLIS was detected by Q-PCR every two months and continuously monitored for 12 months. In the TFR period, the peripheral blood BCR/ABLIS was detected once a month for the first 6 months; the peripheral blood BCR/ABLIS was detected once every two months for the next 6 months; after that, the peripheral blood BCR/ABLIS was detected once every three months.

3.If the patients detected molecular recurrence (loss of MMR, BCR/ABL IS>0.1%),the original dose of 2G-TKI should be administered

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over 18 years
2. Patients diagnosed as Ph+ (or Ph- but PCR-positive for BCR-ABL) CML-CP
3. Patients have received one of the second-generation TKIs (nilotinib, dasatinib) for at least 3 years
4. Patients have maintained MMR (BCR/ABL IS<0.1% or more) at least 2 years
5. in the past 24 months, at least three times recent molecular reactions have confirmed MMR
6. Patients have signed the informed consent

Exclusion Criteria:

1. patients with the presence or history of T315I mutation
2. patients with the presence of rare unquantifiable atypical transcripts
3. Patients with comorbid cardiovascular disease or a history of severe cardiovascular disease
4. patients have history of accelerated or blast phase, or suspected blast disease
5. patients have received allogeneic hematopoietic stem cell transplantation
6. patients have severe abnormal liver and kidney function (ALT > upper limit of normal, AST > 3 times normal upper line, glomerular filtration rate < 50%)
7. patients combined with other tumors or a history of other malignancies ECOG score>3
8. Two-line abnormality in the patient's blood routine examination
9. women is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been diagnosed with CML-CP and are older than 18 years
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
MMR(BCR/ABL IS<0.1%) on 24 months | 24 months
  Continue to treat patients at half-dose for 12 months, then stop for 12 months

SECONDARY OUTCOMES:
MRFS | 24 months
  Molecular relapse free survival in 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- NanfangH, Guangzhou, Guangdong, China